CLINICAL TRIAL: NCT03379493
Title: Open-label Phase I Study of ET190L1 ARTEMIS™ T Cells in Relapsed and Refractory CD19+ Non-Hodgkin's Lymphoma
Brief Title: Study of ET190L1 ARTEMIS™ T Cells in Relapsed and Refractory CD19+ Non-Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor's Decision
Sponsor: Eureka Therapeutics Inc. (Industry)
Collaborators: Duke University (Other); Duke Clinical Research Institute (Other)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ETUS16CD19AR107
Record Dates: First submitted 2017-12-13; First posted 2017-12-20 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Lymphomas Non-Hodgkin's B-Cell
Keywords: relapsed/refractory CD19+ Lymphomas Non-Hodgkin's B-Cell
MeSH Terms: conditions — Lymphoma, B-Cell; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ET190L1 ARTEMIS™ T cells (Experimental): ET190L1 ARTEMIS™ T cells administered by intravenous (IV) infusion
  Interventions: Biological: ET190L1 ARTEMIS™ T cells

INTERVENTIONS:
Biological: ET190L1 ARTEMIS™ T cells — Autologous T cells transduced with lentivirus encoding an anti-CD19 (ET190L1) ARTEMIS™ expression construct, administered by intravenous (IV) infusion

SUMMARY:
This is a non-randomized, single arm, open-label, single institution, phase I study to determine the maximum tolerated dose (MTD) of ET190L1 ARTEMIS™ T cells in patients ≥ 18 years of age with relapsed or refractory CD19+ Non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
The trial will follow a traditional dose-escalation model to establish the MTD and recommended phase 2 dose (RP2D) of infused ET190L1 ARTEMIS™ T cells following lympho-depleting chemotherapy. Two sequential cohorts of patients will be recruited to fulfill this study, those in the dose escalation cohort (for determination of MTD and RP2D) and those in the expansion cohort (treated on the RP2D). The study will have concurrent phases of screening, pre-treatment, treatment, primary follow-up, safety, and survival follow-up. The total duration of the study involvement for the patient is 15 years. Efficacy will be assessed until progression and safety will be assessed throughout the full duration of the study. Twelve to 24 patients will be treated to determine the MTD. Following determination of the MTD, an expansion cohort consisting of 6 patients per disease subtype (n= 30) will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsed/refractory CD19+ Non-Hodgkin's lymphoma of the following subtypes:

  * Diffuse large B-cell lymphoma (DLBCL)
  * Mantle cell lymphoma (MCL)
  * Follicular lymphoma (FL)
  * Chronic lymphocytic leukemia and Small lymphocytic lymphoma (CLL/SLL)
  * Burkitt's Lymphoma
* Ability to provide written informed consent for the protocol.
* Willingness and ability to comply with scheduled visit, treatment plans, laboratory tests, and other procedures.
* Age ≥ 18 years old.
* Eastern Cooperative Oncology Group performance status of ≤ 2.
* Evidence of at least one measurable lesion (nodes/nodal masses > 1.5 cm, extranodal masses >1.0 cm or PET avid lesions consistent with lymphoma) on imaging with the following exceptions:

  1. Patients treated with interim chemotherapy for disease control between enrollment and ET190L1 ARTEMIS™ T cell infusion who do not have measurable disease at re-screening are still eligible.
  2. CLL/SLL with documented B-cell absolute lymphocytosis > 5 x 109 cells/L peripheral blood or infiltration of lymph nodes and/or bone marrow infiltration by CLL phenotype cells defined as: clonal B cells with majority population co-expressing CD5 and CD19, with surface immunoglobulin (sIg, kappa or lambda but not both) and CD20 (dim), CD23+ (if CD20 or sIg are bright or if CD23 is dim or negative [atypical CLL phenotype] then FISH for 11:14 translocation must be performed to differentiate from mantle cell lymphoma).
  3. Lesions previously irradiated will be considered measurable only if progression has been documented following completion of radiation therapy.
* Must have biopsy-proven primary refractory disease or relapsed disease after front-line chemo-immunotherapy (with anti-CD20 mAb in combination with anthracycline-based chemotherapy) or at least one of the following:

  * For subjects with DLBCL: relapsed or refractory disease after ≥ 2 prior line(s) of therapy. For both de novo and transformed disease, patients must have received at least 1 prior regimen with anti-CD20 mAb and anthracycline.
  * For subjects with FL or SLL: relapsed or refractory disease after ≥ 2 prior line(s) of therapy.
  * For subjects with CLL: must be relapsed or refractory disease and:

    1. with no unfavorable cytogenetics and have failed ≥ 3 prior line(s) of therapy.
    2. with unfavorable cytogenetics including del17p/mutated p53 or unmutated immunoglobulin heavy chain variable region relapsed or refractory disease after ≥ 2 prior line(s) of therapy which must have included ibrutinib.
  * For subjects with MCL: relapsed or refractory disease after at least 1 prior regimen with chemoimmunotherapy.
  * For subjects with Burkitt's: relapsed or refractory disease after at least 1 prior line of therapy.
  * Any patient, with subtypes listed above, having either failed autologous HSCT after at least 1 prior regimen, or those patients ineligible for, but not an appropriate candidate, or not consenting to autologous HSCT.
* Adequate organ function parameters are set according to what the treating physician defines as adequate organ function and are acceptable for participation in this trial. These criteria are defined as:

  1. Renal function:

     1. Creatinine clearance ≥45ml/min
  2. Liver function:

     1. AST/ALT ≤ 3x the institutional ULN, except for people with liver involvement by their lymphoma, who may be included if AST/ALT ≤ 5x the institutional ULN.
     2. Total bilirubin ≤ 2x the institutional ULN with the exception of patients with Gilbert syndrome; patients with Gilbert syndrome may be included if their total bilirubin is ≤ 3.0x ULN and direct bilirubin is ≤ 2x ULN
  3. Pulmonary function:

     1. Must have a minimum level of pulmonary reserve defined as ≤ Grade 1 dyspnea and pulse oximetry of ≥ 88% on room air.
  4. Cardiac function:

     1. Must be hemodynamically stable at the time of ET190L1 ARTEMIS™ T cell administration and have LVEF ≥ 45% confirmed by echocardiogram or MUGA scan
  5. Bone marrow reserve without transfusion defined as:

     1. Absolute neutrophil count (ANC) ≥ 1,000/mm3
     2. Absolute lymphocyte count (ALC) ≥ 300/mm3, and absolute number of CD3+ T cells > 150/mm3
     3. Platelets ≥ 50,000/mm3
     4. Hemoglobin ≥ 8 g/dL
* Women who are pregnant will be excluded from the study. A woman of child-bearing potential, defined as all women physiologically capable of becoming pregnant, will have a blood pregnancy test and the test must be negative to participate in this study. Women of child-bearing potential and all male participants must use effective methods of contraception for at least 12 months following infusion of ET190L1 ARTEMIS™ T cells and until ET190L1 ARTEMIS™ T cells are no longer present by PCR (with surveillance to cease at 5 years).

  1. Medically acceptable contraceptives for females include:

     1. Surgical sterilization (such as a tubal ligation or hysterectomy).
     2. Approved hormonal contraceptives (such as birth control pills, patches, implants, or injections).
     3. Barrier methods (such as condoms or diaphragms) used with a spermicide.
     4. An intrauterine device (IUD).
  2. Contraceptive measures such as Plan B, sold for emergency use after unprotected sex, are not acceptable methods for routine use. If the woman does become pregnant during this study or if the woman has unprotected sex, she must inform the study physician immediately.
  3. Medically acceptable contraceptives for males include:

     1. Surgical sterilization (such as a vasectomy)
     2. A condom used with a spermicide
  4. Contraceptive measures such as Plan B, sold for emergency use after unprotected sex, are not acceptable methods for routine use. The man should inform his partner of the potential for harm to an unborn child. She should know that if pregnancy occurs, he will need to report it to the study doctor, and she should promptly notify her doctor.

Exclusion Criteria:

* Prior Treatment:

  1. With any prior anti-CD19/anti-CD19 CAR-T or cellular therapy (prior Blinotumomab therapy is allowed)
  2. Treatment with any prior gene therapy
  3. Prior allogeneic hematopoietic stem cell transplant
  4. Received chemotherapy, radiation or surgical resection of malignancy within 2 weeks prior to the start of conditioning chemotherapy (day -10 to -5).
* Active, uncontrolled serious infection or medical or psychiatric illness, that in the investigator's opinion is likely to interfere with participation in this clinical trial
* Active CNS involvement by malignancy.
* History of seizure disorder, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease with CNS involvement.
* Active replication of hepatitis B or active hepatitis C (HCV RNA positive). Those with prior disease who are PCR negative at enrollment and meet liver function eligibility criterion are eligible.
* Known HIV positive patients
* Patients with unstable angina and/or myocardial infarction within 6 months prior to screening.
* Cardiac arrhythmia not controlled with medical management, evidence of pericardial effusion on imaging that is compromising function.
* Previous or concurrent malignancy with exception of adequately treated basal cell or squamous cell carcinoma, in-situ carcinoma of the cervix or breast, treated curatively and without evidence of recurrence for at least 3 years prior to study drug infusion, or prostate cancer that was treated with prostatectomy or radiotherapy over 2 years before day 1 of protocol therapy and patients whose PSA is undetectable at study entry.
* Autoimmune disease or history of primary immunodeficiency (excluding Hashimoto's thyroiditis, vitiligo, or DM type I)
* Women who are pregnant or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2018-12-23 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 24 months
  Estimate the maximum tolerated dose of ET190L1 ARTEMIS™ T cells in patients with a relapsed and/or refractory CD19+ Non-Hodgkin's lymphoma
Toxicity profile of ET190L1 ARTEMIS™ T-cell treatment | 24 months
  The frequency of occurrence and severity of treatment-related adverse events, including adverse events of special interest (AESI) will be reported. AESI include: CRS (severity grade 1-5), Tumor Lysis Syndrome, Neutropenic Fever, Cytopenia lasting >28 days, neurotoxicity (severity grade 1-5), hypogammaglobulinemia and reductions in cardiac function.

SECONDARY OUTCOMES:
Overall response rate (ORR) | 24 months
  Evaluate the efficacy of ET190L1 ARTEMIS™ T cell therapy, defined as overall response rate (ORR), including CR or PR, of patients with relapsed/refractory CD19+ Non-Hodgkin's lymphoma who receive human ET190L1 ARTEMIS™ T cell therapy. Evaluation, staging and response assessment will be carried out using the Lugano classification
Overall response rate (ORR) in histologic subtypes of CD19+ Non-Hodgkin's lymphoma | 24 months
  Evaluate the efficacy of ET190L1 ARTEMIS™ T cells in histologic subtypes of CD19+ Non-Hodgkin's lymphoma.
Duration of overall response (DOR) | 24 months
  Evaluate duration of overall response (DOR)
Progression free survival (PFS) | 24 months
  Evaluate progression free survival (PFS)
Overall survival (OS) | 24 months
  Evaluate overall survival (OS)

CONTACTS AND LOCATIONS:
Overall Officials: David A Rizzieri, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No